CLINICAL TRIAL: NCT07137325
Title: Investigating the Effects of Play Therapy Techniques on Learned Helplessness and Social Comparison Levels in Children Living in an Orphanage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Principal Investigator, Fatih Sahin, principal investigator, Muş Alparslan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 134665
Record Dates: First submitted 2025-07-31; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2024-08

CONDITIONS: Learned Helplessness; Social Comparison
MeSH Terms: interventions — Play Therapy

STUDY DESIGN:
Intervention Model Description: The data collection process consisted of three stages. In the first stage, pretest data were collected by administering the Learned Helplessness Scale and the Social Comparison Scale to both groups before the intervention. In the second stage, structured play therapy sessions, each approximately 60 minutes long, were administered to the children in the experimental group once a week for six weeks. These sessions consisted of play therapy techniques focusing on developmental appropriateness, emotional expression, problem solving, and self-perception. The control group received no intervention during this period. In the third stage, after the intervention was completed, the same scales were administered to both groups again to obtain posttest data. The data collection process lasted a total of six weeks, and the sessions were conducted one-on-one in appropriate, quiet, and safe environments in the children's homes. All sessions were conducted by the researcher, and the principle of volun
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Play therapy techniques were applied for 6 weeks.
  Interventions: Behavioral: play therapy
- control group (No Intervention): no intervention was implemented

INTERVENTIONS:
Behavioral: play therapy — The intervention consisted of a structured play therapy program specifically designed for children residing in institutional care settings. What distinguishes this intervention from others is its targeted focus on reducing learned helplessness and improving social comparison tendencies, two psychological constructs particularly relevant to children in residential care.
  The program was conducted over six weekly sessions, each lasting approximately 60 minutes, and implemented in a one-on-one format within a safe, quiet room in the child care facility. The content was developmentally appropriate and included modules on emotional expression, communication, realistic goal setting, resource awareness, problem-solving, and positive self-perception. The therapeutic techniques were based on principles of non-directive and humanistic play therapy, allowing children to express themselves freely while being guided through structured themes.
  Unlike general play therapy programs, this intervention
  Arms: experimental group

SUMMARY:
Purpose: This study aims to examine the effects of play therapy techniques on the learned helplessness levels and social comparison tendencies of children living in children's homes.

DETAILED DESCRIPTION:
Purpose: This study aims to examine the effects of play therapy techniques on the learned helplessness levels and social comparison tendencies of children living in children's homes.

Method: The study was conducted using a randomized experimental design with a pretest-posttest control group. The research sample consisted of 39 children living in children's homes affiliated with the Ministry of Family and Social Services in Türkiye. Participants were randomly assigned to experimental (n=21) and control (n=18) groups. The experimental group received a six-week structured play therapy program. Data were collected using a Personal Information Form, the Learned Helplessness Scale, and the Social Comparison Scale, and nonparametric tests were used in analyses.

ELIGIBILITY:
Inclusion Criteria:

* - Living in a children's home,
* Continuing education,
* Having no hearing or vision problems.

Exclusion Criteria:

* those who do not meet the inclusion criteria

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
pretest (6-week play therapy before the intervention) | Baseline (within 1 week before play therapy)
  Primary Outcome Measure 1: Social Comparison Level (Social Comparison Scale)
  Description: Social Comparison Scale, range 12-60; higher scores = higher social comparison tendency.
  Time Frame: Baseline (pre-intervention, within 1 week before play therapy).
  Unit of Measure: Total score (12-60).
pretest (6-week play therapy before the intervention) | Time Frame: Baseline (pre-intervention, within 1 week before play therapy).
  Primary Outcome Measure 2: Learned Helplessness Level (Learned Helplessness Scale)
  Description: Learned Helplessness Scale, range 0-20; higher scores = greater learned helplessness.
  Time Frame: Baseline (pre-intervention, within 1 week before play therapy).
  Unit of Measure: Total score (0-20).

SECONDARY OUTCOMES:
posttest (After the 6-week play therapy intervention) | At 6 weeks (immediately after completion of play therapy).
  Secondary Outcome Measure 1: Social Comparison Level Post-Intervention (Social Comparison Scale)
  Description: Social Comparison Scale, range 12-60; higher scores = higher social comparison tendency.
  Time Frame: Post-intervention (at 6 weeks after completion of play therapy).
  Unit of Measure: Total score (12-60).
posttest (After the 6-week play therapy intervention) | 6 weeks after baseline (post-intervention)
  Secondary Outcome Measure 2: Learned Helplessness Level Post-Intervention (Learned Helplessness Scale)
  Description: Learned Helplessness Scale, range 0-20; higher scores = greater learned helplessness.
  Time Frame: Post-intervention (at 6 weeks after completion of play therapy).
  Unit of Measure: Total score (0-20).

CONTACTS AND LOCATIONS:
Locations (1):
- Aile Ve Sosyal Hizmetler Il Müdürlüğü, Muş, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) will not be made publicly available but may be shared upon reasonable request. Data sharing will be considered on a case-by-case basis and only for academic, non-commercial purposes. Sharing will be subject to legal and ethical restrictions, including the protection of participant confidentiality and compliance with institutional ethics approval.